CLINICAL TRIAL: NCT03815981
Title: Linking Iron-deficiency With Allergy- the Role of Microbial Survival Components
Brief Title: Siderophore-profile in Allergic and Non-allergic Subjects
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Franziska Roth-Walter, Principal Investigator, Medical University of Vienna
Other Study IDs: 1972/2017
Record Dates: First submitted 2019-01-21; First posted 2019-01-25 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Allergy; Healthy; Allergic Sensitisation
Keywords: iron; siderophores; allergy; allergic sensitisation; trace elements
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood, Stool, Urin samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Allergic: Collection of blood, stool, urin samples
- Sensitized: Collection of blood, stool, urin samples
- Non-Allergic: Collection of blood, stool, urin samples

SUMMARY:
This study aims to profile the siderophore-content in the human gut from allergic and non-allergic subjects and to assess their contribution in iron homeostasis.

DETAILED DESCRIPTION:
Iron is an essential nutrient for the majority of commensal bacteria, which commonly secrete siderophores to liberate iron from their surroundings. In several studies, a misbalanced microbiota has been demonstrated in allergics suggesting that also their siderophore profile is severely attenuated.

There are currently no data and very limited knowledge present on the composition of bacterial surviving factors in humans, or on their impact on the human immune system.

As such, 1) the iron status, 2) the microbial biota composition and the 3) siderophore-profile in allergics and non-allergics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* allergic and non-allergic volunteers

Exclusion Criteria:

* Patients will not be considered for the study if they have co-morbidities such as diabetes mellitus, disorders of the liver including hemochromatosis or kidney, autoimmune or metabolic diseases and malignancy or if they use of medications (e.g. antibiotics, PPIs) that influence the iron, inflammatory or microbial status. Further exclusion criteria are pregnancy, lactation; veganism, zinc, and iron supplementation and smoking. Volunteers will be asked to cease blood donation for at least three months' before recruitment and to cease other supplements for at least two weeks, e.g. vitamins, fish oil or minerals (other than zinc and iron).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Allergics and Non-Allergic subjects over 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Iron status | baseline
  Hemoglobin, Ferritin, hepcidin, iron and soluble transferrin receptor concentrations, transferrin saturation in %

SECONDARY OUTCOMES:
Siderophore profile | baseline
  Mass spectrometric analysis of siderophores

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Roth-Walter, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roth-Walter F, Pacios LF, Bianchini R, Jensen-Jarolim E. Linking iron-deficiency with allergy: role of molecular allergens and the microbiome. Metallomics. 2017 Dec 1;9(12):1676-1692. doi: 10.1039/c7mt00241f. Epub 2017 Nov 9. PMID 29120476
- [Derived] Petje LM, Jensen SA, Szikora S, Sulzbacher M, Bartosik T, Pjevac P, Hausmann B, Hufnagl K, Untersmayr E, Fischer L, Vyskocil E, Eckl-Dorna J, Jensen-Jarolim E, Hofstetter G, Afify SM, Krenn CG, Roth GA, Rivelles E, Hann S, Roth-Walter F. Functional iron-deficiency in women with allergic rhinitis is associated with symptoms after nasal provocation and lack of iron-sequestering microbes. Allergy. 2021 Sep;76(9):2882-2886. doi: 10.1111/all.14960. Epub 2021 Jun 17. No abstract available. PMID 34037999